CLINICAL TRIAL: NCT01137045
Title: An Immunogenicity and Safety Study of Modified TRC-ID Regimen With A New Chromatographically Purified Vero Cell Rabies Vaccine(SPEEDA/TRCS SPEEDA) and Rabies Immunoglobulin
Brief Title: Immunogenicity and Safety Study of A New Chromatographically Purified Vero Cell Rabies Vaccine With ID Regimen and ERIG
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Queen Saovabha Memorial Institute (Other)
Responsible Party: Principal Investigator, Suda Sibunruang, Principal investigator, Queen Saovabha Memorial Institute
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: RC5301
Record Dates: First submitted 2010-06-03; First posted 2010-06-04 (Estimated); Last update posted 2018-04-06 (Actual); Status verified 2018-04

CONDITIONS: Rabies
Keywords: rabies vaccine; vero cells; serology; safety
MeSH Terms: conditions — Rabies

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- SPEEDA with modified TRC-ID regimen (Active Comparator): 35 healthy volunteers
  Interventions: Biological: SPEEDA and TRCS SPEEDA
- VERORAB with modified TRC-ID regimen (Active Comparator): 35 healthy volunteers
  Interventions: Biological: SPEEDA and TRCS SPEEDA
- SPEEDA with modified TRC-ID regimen plus ERIG (Active Comparator): 35 healthy volunteers
  Interventions: Biological: SPEEDA and TRCS SPEEDA
- VERORAB with modified TRC-ID regimen plus ERIG (Active Comparator): 35 WHO category III patients
  Interventions: Biological: SPEEDA and TRCS SPEEDA
- SPEEDA with ESSEN IM regimen plus ERIG (Active Comparator): 35 healthy volunteers
  Interventions: Biological: SPEEDA and TRCS SPEEDA
- TRCS SPEEDA with modified TRC-ID regimen plus ERIG (Active Comparator): 35 healthy volunteers
  Interventions: Biological: SPEEDA and TRCS SPEEDA

INTERVENTIONS:
Biological: SPEEDA and TRCS SPEEDA — For modified TRC-ID regimen,0.1 ml of SPEEDA, TRCS SPEEDA or VERORAB will be given at each of two sites,intradermally on upper arms on days 0,3,7 and 28.
  For ESSEN regimen, 1 vial of SPEEDA will be given intramuscularly at upper arm on days 0,3,7,14 and 28.
  For ERIG,it would be given in a single dose 40 IU/Kg at the same time as the first dose of vaccine. ERIG will be infiltrated around and into all wounds as recommended by WHO for patients in group IV and injected intramuscular at each of both gluteal areas for participants in group III,V,VI
  Other Names: SPEEDA; TRCS SPEEDA

SUMMARY:
A comparative,randomized (1:1)study to evaluate the safety and immunogenicity of a new chromatographically purified vero cell rabies vaccine (SPEEDA) and chromatographically purified vero cell rabies vaccine (SPEEDA)which is filled by Queen Saovabha Memorial Institute (TRCS SPEEDA)vs. reference vaccine (purified vero cell vaccine; VERORAB)when using with post-exposure rabies intradermal vaccination with or without equine rabies immunoglobulin.

DETAILED DESCRIPTION:
Rabies is an important world health problem especially in developing countries.Although the case-fatality ratio of human rabies is 100%,the disease is preventable by the modern cell-culture vaccine and rabies immunoglobulin.Post-exposure rabies vaccination with the modified Thai Red Cross intradermal(modified TRC-ID)regimen has been approved by WHO and proven to be immunogenic and effective. It represents a significant saving in vaccine cost and is now established in several developing countries. SPEEDA,chromatography purified vero cell derived rabies vaccine,approved by Thai FDA on 8 April 2009 and drug registration code of SPEEDA is 1C 90022/51. This study has a goal to determine the immunogenicity and safety of SPEEDA and TRCS-SPEEDA (SPEEDA which is filled by Queen Saovabha Memorial Institute)vs. reference vaccine (purified vero cell vaccine; VERORAB)when using with post-exposure rabies intradermal vaccination with or without equine rabies immunoglobulin.

ELIGIBILITY:
Inclusion Criteria:

* subjects are healthy population older than 15 years.
* subjects are willing to give signed informed consents.
* subjects are willing to give blood samples on recommended days.
* subjects are available for follow up according to the table of administration

Exclusion Criteria:

* subjects who had received any type of rabies vaccination in the past
* subjects who had received rabies immunoglobulin in the past
* subjects who had known as immunocompromised hosts
* subjects on steroids or any other immunosuppressant
* subjects on concomitant antimalarials
* subjects who have received of any blood products within the previous 3 months
* subjects with history of allergy to any ingredient of the vaccine
* subjects who had known as pregnancy in first recruitment

Ages: 15 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 210 (Actual)
Dates: Start 2010-06; Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
immunogenicity (the level of rabies neutralizing antibodies by RFFIT test) | 32 months
  The immunogenicity (Rabies neutralizing antibodies) would be checked from the blood samples for 7 times (on days 0,7,14,28,90,180 and 360)for one year duration in each phase.

SECONDARY OUTCOMES:
safety | 32 months
  This would based on general examination, local examination and subjective evaluation of both solicited and unsolicited adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Terapong Tantawichien, MD.,Prof, Principal Investigator — Queen Saovabha Memorial Institute
Locations (2):
- Thailand (2):
  - Suda Sibunruang, Bangkok
  - Queen Saovabha Memorial Institute, Bangkok